CLINICAL TRIAL: NCT07082270
Title: Phase I Trial of GB1211 (Selvigaltin), an Oral Galectin-3 (Gal-3) Inhibitor, Combined With Standard of Care Treatment in Relapsed/Refractory Multiple Myeloma (RRMM)
Brief Title: Selvigaltin With Standard of Care Treatment for the Treatment of Relapsed/Refractory Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-4514825; NCI-2025-04757 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-4514825 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Specimen Handling; Biopsy; carfilzomib; daratumumab; Hyaluronoglucosaminidase; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (selvigaltin, Dara-KD) (Experimental): See Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Carfilzomib; Procedure: Computed Tomography; Drug: Daratumumab and Recombinant Human Hyaluronidase; Drug: Dexamethasone; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Selvigaltin

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Carfilzomib — Given IV
  Other Names: Carfilnat; CFZ; Kyprolis; PR 171; PR-171; PR171
Procedure: Computed Tomography — Undergo PET/CT and/or CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Daratumumab and Recombinant Human Hyaluronidase — Given SC
  Other Names: DARA Co-formulated with rHuPH20; DARA/rHuPH20; Daratumumab + rHuPH20; Daratumumab and Hyaluronidase; Daratumumab and Hyaluronidase-fihj; Daratumumab and vorhyaluronidase; Daratumumab and Vorhyaluronidase Alfa; Daratumumab with rHuPH20; Daratumumab-rHuPH20; Daratumumab/Hyaluronidase-fihj; Daratumumab/rHuPH20 Co-formulation; Darzalex Faspro; Darzalex/rHuPH20; Darzquro; HuMax-CD38-rHuPH20; Recombinant Human Hyaluronidase Mixed with Daratumumab
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Drug: Selvigaltin — Given PO

SUMMARY:
This phase I trial studies the side effects and best dose of selvigaltin when given together with standard of care treatment (daratumumab-hyaluronidase, carfilzomib, dexamethasone) in treating patients with multiple myeloma that has come back after a period of improvement (relapsed) or that does not respond to treatment (refractory). Selvigaltin works by blocking the activity of a protein called galectin-3. Galectin-3 is involved in various cellular processes, including inflammation and tissue scarring, which is associated with worse outcomes in several forms of cancer. By blocking the activity of galectin-3, selvigaltin may help reduce inflammation and tissue scarring. Daratumumab-hyaluronidase is a drug composed of daratumumab and hyaluronidase. Daratumumab is in a class of medications called monoclonal antibodies. It binds to a protein called CD38, which is found on some types of immune cells and cancer cells, including myeloma cells. Daratumumab may block CD38 and help the immune system kill cancer cells. Hyaluronidase helps deliver the daratumumab to CD38-expressing cancer cells. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Dexamethasone is in a class of medications called corticosteroids. It is used to reduce inflammation and lower the body's immune response to help lessen the side effects of chemotherapy drugs. Giving selvigaltin with standard of care treatment may be safe, tolerable, and/or effective in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of selvigaltin in combination with standard of care treatment regimen (daratumumab, carfilzomib, and dexamethasone) for relapsed/refractory multiple myeloma (RRMM).

II. Determine the maximal tolerated dose (MTD) of selvigaltin in combination with a standard of care treatment regimen (daratumumab, carfilzomib, and dexamethasone) for RRMM.

SECONDARY OBJECTIVES:

I. To collect safety and preliminary efficacy data. II. Rate of bone marrow measurable residual disease (MRD) negativity.

EXPLORATORY OBJECTIVE:

I. To assess the effects of the combination treatment on the tumor microenvironment (TME) and on immune cell subsets in the peripheral blood and bone marrow.

OUTLINE: This is a dose-escalation study of selvigaltin in combination with daratumumab and recombinant human hyaluronidase (daratumumab-hyaluronidase), carfilzomib, and dexamethasone followed by a dose-expansion study.

Patients receive selvigaltin orally (PO) twice daily (BID) on days 1-28 of each cycle, daratumumab-hyaluronidase subcutaneously (SC) on days 1, 8, 15, and 22 of cycles 1-2 and days 1 and 15 of cycles 3-6, carfilzomib intravenously (IV) over 30 minutes on days 1, 8, and 15 of each cycle, and dexamethasone PO on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients who respond to treatment may optionally continue to receive treatment beyond 6 cycles with selvigaltin PO BID on days 1-28 of each cycle, daratumumab-hyaluronidase SC on day 1 of each cycle, carfilzomib IV over 30 minutes on days 1, 8, and 15 of each cycle, and dexamethasone PO on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening and blood sample collection and bone marrow aspiration and biopsy throughout the trial. Patients also undergo positron emission tomography (PET)/computed tomography (CT), magnetic resonance imaging (MRI), and/or CT during screening and optionally during 1 year follow up.

After completion of study treatment, patients that remain on treatment beyond 6 cycles are followed up monthly until disease progression and then every 3 months for up to 3 years. Patients that do not continue treatment are followed up at 30 days and then every 3 months for up to 3 years or until start of a new treatment, disease progression, or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* RRMM with measurable disease prior to initiation of study intervention. Measurable disease must include at least one of the following criteria:

  * Serum M-protein > 0.5 g/dL or,
  * Urine M-protein > 200 mg/24h or,
  * Serum free light chain assay: involved free light chain (FLC) level > 100 mg/L provided serum free light chain ratio is abnormal or,
  * Bone marrow plasma cells > 10% of total bone marrow cells
* Have received ≥ 1 prior line of therapy
* Planned treatment with the standard of care regimen of daratumumab, carfilzomib, and dexamethasone (Dara-KD) regimen
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Absolute neutrophil count: ≥ 1,000 /µL
* Platelets: ≥ 75,000 /µL
* Hemoglobin: ≥ 7 g/dL
* Total bilirubin: ≤ 1.5 x upper limit of normal (ULN): ≤ 3.0 x ULN for Gilbert's Syndrome
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]): ≤ 3 x ULN
* Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min
* Left ventricular ejection fraction of at least 50% by ECHO or MUGA
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for 6 months following the last dose of the investigational drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participants must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Known hypersensitivity to selvigaltin or any of the excipients
* Prior hypersensitivity or grade 3 skin toxicity with daratumumab/carfilzomib
* Exposure to prior daratumumab/carfilzomib is permitted, however refractoriness within 6 months of study initiation is exclusionary
* Concomitant medication(s) known to be (a) a strong inhibitor or inducer of CYP3A4, (b) strong P-gp/MDRI inhibitors or inducers or, (c) QT interval (QT) prolonging as defined in the drug's label, with the exception of drugs that are considered absolutely essential for the care of the subject or if the Investigator believes that beginning therapy with such medication is vital to an individual subject's care while on study, and in either case, there is no alternative medication
* Electrocardiogram (ECG) demonstrating a corrected QT interval (QTc) interval > 470 msec without a bundle block or patients with congenital long QT syndrome
* Coronary artery bypass, angioplasty, vascular stent, myocardial infarction, angina or congestive heart failure in the last 6 months
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, class III or IV heart failure (New York Heart Association functional classification system), or psychiatric illness/social situations that would limit compliance with study requirements
* Known active bacillus tuberculosis infection
* Known active HIV unless CD4+ > 350 cells/µL, no history of AIDS-defining opportunistic infection within the past 12 months, or on effect anti-retroviral therapy (ART) with > 4 weeks on treatment and viral load < 400 copies/mL. Confirm low risk of drug-drug interactions or are able to be substituted
* Pregnant or nursing female participants
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | Up to 28 days
  As assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version (v) 5.0. The DLTs will be summarized by dose level using frequencies and relative frequencies.
Maximum tolerated dose (MTD) | Up to 28 days
  Will determine the MTD of selvigaltin when administered in combination with daratumumab, carfilzomib, and dexamethasone (DaraKD). Will employ the Bayesian optimal interval design to find the MTD.
Recommended phase 2 dose (RP2D) | Up to 28 days
  Will determine the RP2D of selvigaltin when administered in combination with DaraKD. The RP2D will be determined by evaluating both the toxicity profile and the therapeutic response.

SECONDARY OUTCOMES:
Incidence of overall adverse events | Up to 6 cycles (Cycle length = 28 days)
  As assessed by the NCI CTCAE v5.0.
Incidence of serious adverse events | Up to 6 cycles (Cycle length = 28 days)
  As assessed by the NCI CTCAE v5.0.
Overall response rate | During or after 6 cycles of therapy, assessed up to 3 years (Cycle length = 28 days)
  As per investigator's assessment using the International Myeloma Working Group criteria will be summarized as proportions and 90% Clopper-Pearson confidence intervals by dose levels.
Duration of response | During or after 6 cycles of therapy, assessed up to 3 years (Cycle length = 28 days)
Progression free survival | From the start of treatment until the first occurrence of disease progression or death from any cause, whichever comes first, assessed up to 3 years
  Will be summarized using Kaplan-Meier estimators by dose levels.
Overall survival | From the start of treatment to death from any cause, assessed up to 3 years
  Will be summarized using Kaplan-Meier estimators by dose levels.
Patient reported outcomes | At baseline, cycle 4 day 1, and 30 days after last dose of study drug
  As assessed using the European Organization for the Research and Treatment of Cancer Quality of Life-Core 30 questionnaire. Will be summarized by dose levels and time points. Generalized linear mixed models will be used for within-subject comparisons between time points.
Bone marrow measurable residual disease (MRD) status | After 6 cycles (Cycle length = 28 days)
  The MRD status will be summarized as frequencies and relative frequencies by dose levels.

CONTACTS AND LOCATIONS:
Overall Officials: Hamza Hassan, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States